CLINICAL TRIAL: NCT04170621
Title: PersAFOne: Feasibility Study of the FARAPULSE™ Endocardial Ablation System in the Treatment of Persistent Atrial Fibrillation
Brief Title: Feasibility Study of the FARAPULSE Endocardial Multi Ablation System in the Treatment of Persistent Atrial Fibrillation
Acronym: PersAFOne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0607
Record Dates: First submitted 2019-10-17; First posted 2019-11-20 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-11

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- FARAPULSE Endocardial Ablation (Experimental): Ablation using the FARAPULSE Endocardial Multi Ablation System
  Interventions: Device: Ablation

INTERVENTIONS:
Device: Ablation — Ablation using the FARAPULSE Endocardial Multi Ablation System

SUMMARY:
PersAFOne:

Feasibility Study of the FARAPULSE™ Endocardial Ablation System in the Treatment of Persistent Atrial Fibrillation

DETAILED DESCRIPTION:
This is a prospective, multi-center safety and feasibility study in subjects with persistent AF. Subjects will undergo percutaneous PEF ablation for pulmonary vein isolation as well as cavotricuspid isthmus interruption and other left atrial ablations at the investigator's discretion. Subjects will then be followed at 30 days, 75 ± 15 days, 6 months and 12 months for adverse events, recurrence of arrhythmia after a 90 day blanking period and other relevant outcome measures.

ELIGIBILITY:
Inclusion Criteria:

Study subjects are required to meet all the following inclusion criteria to participate in this study:

1. Patients with documented drug-resistant symptomatic persistent AF meeting all three of the following criteria:

   1. Patient is refractory or intolerant to at least one Class I/III antiarrhythmic agent.
   2. ECG-documented first episode of persistent AF, lasting longer than 7 days but not longer than 365 days
   3. Holter within 90 days of the Enrollment Date demonstrating 24 hours of continuous AF
2. Patients who are ≥ 18 and ≤ 75 years of age on the day of enrollment.
3. Patient participation requirements:

   1. Lives locally
   2. Is willing and capable of providing Informed Consent to undergo study procedures
   3. Is willing to participate in all examinations and follow-up visits and tests associated with this clinical study.

Exclusion Criteria:

Subjects will be excluded from participating in this study if they meet any one of the following exclusion criteria:

1. AF that is:

   1. Paroxysmal (longest AF episode < 7days)
   2. Longstanding (has persisted > 12 months or that does not respond to cardioversion if < 12 months)
   3. Secondary to electrolyte imbalance, thyroid disease, alcohol abuse or other reversible / non-cardiac causes
2. Left atrial anteroposterior diameter ≥ 5.5 cm as documented by transthoracic echocardiography (TTE) or computed tomography (CT)
3. Any of the following cardiac procedures, implants or conditions:

   1. Clinically significant arrhythmias other than AF, AFL or AT
   2. Hemodynamically significant valvular disease
   3. Prosthetic heart valve
   4. NYHA Class III or IV CHF
   5. Previous endocardial or epicardial ablation or surgery for AF
   6. Atrial or ventricular septal defect closure
   7. Atrial myxoma
   8. Left atrial appendage device or occlusion
   9. Pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy devices
   10. Significant or symptomatic hypotension
   11. Bradycardia or chronotropic incompetence
   12. History of pericarditis
   13. History of rheumatic fever
   14. History of congenital heart disease with any residual anatomic or conduction abnormality
4. Any of the following within 3 months of enrollment:

   1. Myocardial infarction
   2. Unstable angina
   3. Percutaneous coronary intervention
   4. Heart surgery (e.g. coronary artery bypass grafting, ventriculotomy, atriotomy)
   5. Heart failure hospitalization
   6. Stroke or TIA
   7. Clinically significant bleeding
   8. Pericarditis or pericardial effusion
   9. Left atrial thrombus
5. History of blood clotting or bleeding abnormalities.
6. Contraindication to, or unwillingness to use, systemic anticoagulation
7. Contraindications to CT or MRI
8. Sensitivity to contrast media not controlled by premedication
9. Women of childbearing potential who are pregnant, lactating or not using birth control
10. Medical conditions that would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or confound data or its interpretation, including but not limited to

    1. Body mass index (BMI) > 40
    2. Solid organ or hematologic transplant, or currently being evaluated for an organ transplant
    3. Severe lung disease, pulmonary hypertension, or any lung disease involving abnormal blood gases or significant dyspnea
    4. Renal insufficiency with an estimated creatinine clearance < 30 mL/min/1.73 m2, or any history of renal dialysis or renal transplant
    5. Active malignancy or history of treated cancer within 24 months of enrollment
    6. Clinically significant gastrointestinal problems involving the esophagus, stomach and/or untreated acid reflux
    7. Clinically significant infection
    8. Predicted life expectancy less than one year
11. Clinically significant psychological condition that in the investigator's opinion would prohibit the subject's ability to meet the protocol requirements
12. Current or anticipated enrollment in any other clinical study
13. Employment by FARAPULSE or the same hospital department or office of any investigator, or a family member of any of the preceding groups.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospital of Split, Split, Croatia
- Nemocnice Na Homolce, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reddy VY, Anic A, Koruth J, Petru J, Funasako M, Minami K, Breskovic T, Sikiric I, Dukkipati SR, Kawamura I, Neuzil P. Pulsed Field Ablation in Patients With Persistent Atrial Fibrillation. J Am Coll Cardiol. 2020 Sep 1;76(9):1068-1080. doi: 10.1016/j.jacc.2020.07.007. PMID 32854842

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FARAPULSE Endocardial Ablation
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FARAPULSE Endocardial Ablation
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Czechia | 16
  Croatia | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety at 30 Days
Description: Occurrence of primary safety events at 30 days post procedure: death, MI, stroke/TIA, thromboembolism, pericarditis/tamponade, vascular access complications, hospitalization, heart block, PV stenosis, atriosesphageal fistula
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE Endocardial Ablation
Number analyzed (Participants) | 28
Participants | 1

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | FARAPULSE Endocardial Ablation
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 4/28
Other Adverse Events (participants affected / at risk) | 13/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE Endocardial Ablation (N=28)
Cataract traumatic (Injury, poisoning and procedural complications) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Corneal Erosion (Eye disorders) | 1 (1)
Tonsilitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE Endocardial Ablation (N=28)
Chronic Gastritis (Gastrointestinal disorders) | 3 (3)
Hiatus Hernia (Gastrointestinal disorders) | 2 (2)
Gastric Disorder (Gastrointestinal disorders) | 1 (1)
Intestinal Metaplasia (Gastrointestinal disorders) | 1 (1)
Hematoma (Vascular disorders) | 2 (2)
Epistaxis (Vascular disorders) | 1 (1)
Vein Disorder (Vascular disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
AV Block 2nd Degree (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Chest Discomfort (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT04170621/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT04170621/SAP_001.pdf